CLINICAL TRIAL: NCT02542293
Title: A Phase III Randomized, Open-Label, Multi-Center, Global Study of MEDI4736 in Combination With Tremelimumab Therapy Versus Standard of Care Platinum-Based Chemotherapy in First-Line Treatment of Patients With Advanced or Metastatic Non Small-Cell Lung Cancer (NSCLC).
Brief Title: Study of Durvalumab With Tremelimumab Versus SoC as 1st Line Therapy in Metastatic Non Small-Cell Lung Cancer (NSCLC) (NEPTUNE)
Acronym: NEPTUNE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419AC00003; 2015-002197-21 (EudraCT Number)
Record Dates: First submitted 2015-08-26; First posted 2015-09-07 (Estimated); Results first posted 2022-05-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Carcinoma NSCLC
Keywords: NSCLC; PDL1; TMB; MEDI4736; Durvalumab; Tremelimumab; OS
MeSH Terms: interventions — CP protocol; Gemcitabine; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination Therapy (Experimental): Durvalumab (PD-L1 monoclonal antibody) + Tremelimumab (monoclonal antibody directed against CTLA-4)
  Interventions: Biological: Durvalumab +Tremelimumab
- Standard of Care (Active Comparator): Standard of Care chemotherapy treatment
  Interventions: Drug: Paclitaxel + carboplatin; Drug: Gemcitabine + cisplatin; Drug: Gemcitabine + carboplatin; Drug: Pemetrexed + cisplatin; Drug: Pemetrexed + carboplatin

INTERVENTIONS:
Biological: Durvalumab +Tremelimumab
  Arms: Combination Therapy
Drug: Paclitaxel + carboplatin — Chemotherapy Agents
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Standard of Care
Drug: Gemcitabine + cisplatin — Chemotherapy Agents
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Standard of Care
Drug: Gemcitabine + carboplatin — Chemotherapy Agents
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Standard of Care
Drug: Pemetrexed + cisplatin — Chemotherapy Agent
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Standard of Care
Drug: Pemetrexed + carboplatin — Chemotherapy Agent
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Standard of Care

SUMMARY:
This is a randomized, open-label, multi-center, global, Phase III study to determine the efficacy and safety of durvalumab + tremelimumab combination therapy versus platinum-based SoC chemotherapy in the first-line treatment of patients with epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) wild-type advanced or metastatic NSCLC.

DETAILED DESCRIPTION:
Patients will be randomized in a 1:1 to receive treatment with durvalumab + tremelimumab combination therapy or SoC therapy. The primary objective of this study is to assess the efficacy of combination treatment compared with SoC in terms of Overall Survival (OS) in patients.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients should fulfill the following criteria:

* Aged at least 18 years
* Documented evidence of Stage IV NSCLC
* No activating EGFR mutation or ALK rearrangement
* No prior chemotherapy or any other systemic therapy for recurrent/metastatic NSCLC
* World Health Organization (WHO) Performance Status of 0 or 1
* No Prior exposure to Immune Mediated Therapy (IMT), including, but not limited to, other antiCTLA4, antiPD1, anti PDL1,or antiPDL2 antibodies, excluding therapeutic anticancer vaccines

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

* Mixed small cell lung cancer and NSCLC histology, sarcomatoid variant
* Brain metastases or spinal cord compression unless the patient is stable (asymptomatic; no evidence of new or emerging brain metastases) and off steroids for at least 14 days prior to start of study treatment.
* Active or prior documented autoimmune or inflammatory disorders (e.g., Crohn's disease, ulcerative colitis)

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 953 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto de Castro, Principal Investigator — Faculdade de Medicina da Universidade de São Paulo
Locations (161):
- United States (15):
  - Research Site, Anaheim, California
  - Research Site, San Diego, California
  - Research Site, Santa Rosa, California
  - Research Site, Louisville, Kentucky
  - Research Site, Florham Park, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, East Setauket, New York
  - Research Site, Fresh Meadows, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Stony Brook, New York
  - Research Site, Canton, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Zanesville, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Houston, Texas
- Argentina (8):
  - Research Site, Berazategui
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Rioja
  - Research Site, Rosario
  - Research Site, San Salvador de Jujuy
  - Research Site, Santa Rosa
- Brazil (8):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Fortaleza
  - Research Site, Ijuí
  - Research Site, Itajaí
  - Research Site, Porto Alegre
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (5):
  - Research Site, Plovdiv
  - Research Site, Shumen
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Vratsa
- Chile (3):
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (8):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Shanghai
  - Research Site, Ürümqi
  - Research Site, Wuhan
- Research Site, Odense C, Denmark
- Finland (2):
  - Research Site, Oulu
  - Research Site, Tampere
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Holargos, Athens
  - Research Site, Ioannina
- Hong Kong (3):
  - Research Site, Hong Kong
  - Research Site, King's Park
  - Research Site, Shatin
- India (6):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Chennai
  - Research Site, Gūrgaon
  - Research Site, Karamsad
  - Research Site, New Delhi
- Israel (6):
  - Research Site, Beersheba
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Nahariya
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
- Japan (25):
  - Research Site, Bunkyō City
  - Research Site, Fukushima
  - Research Site, Habikino-shi
  - Research Site, Hirosaki-shi
  - Research Site, Iizuka-shi
  - Research Site, Iwakuni-shi
  - Research Site, Kanazawa
  - Research Site, Kishiwada-shi
  - Research Site, Kobe
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Mitaka-shi
  - Research Site, Nagaoka-shi
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Saga
  - Research Site, Sagamihara-shi
  - Research Site, Sakaishi
  - Research Site, Sendai
  - Research Site, Tokushima
  - Research Site, Ube-shi
  - Research Site, Wakayama
  - Research Site, Yokohama
- Malaysia (3):
  - Research Site, Kuala Lumpur
  - Research Site, Kuantan
  - Research Site, Kuching
- Mexico (5):
  - Research Site, Acapulco
  - Research Site, Aguascalientes
  - Research Site, Mérida
  - Research Site, México
  - Research Site, Monterrey
- Peru (3):
  - Research Site, Arequipa
  - Research Site, Bellavista
  - Research Site, Lima
- Philippines (5):
  - Research Site, Baguio City
  - Research Site, Cebu
  - Research Site, Las Piñas
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (9):
  - Research Site, Bydgoszcz
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Mrozy
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wodzisław Śląski
- Portugal (3):
  - Research Site, Amadora
  - Research Site, Lisbon
  - Research Site, Porto
- Research Site, Doha, Qatar
- Research Site, Suceava, Romania
- Russia (3):
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Saint Petersburg
- Saudi Arabia (2):
  - Research Site, Dammam
  - Research Site, Riyadh
- Research Site, Singapore, Singapore
- South Korea (3):
  - Research Site, Daegu
  - Research Site, Hwasun-gun
  - Research Site, Seoul
- Sweden (4):
  - Research Site, Eskilstuna
  - Research Site, Linköping
  - Research Site, Stockholm
  - Research Site, Uppsala
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
- Ukraine (13):
  - Research Site, Chernivtsі
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kapitanivka Village
  - Research Site, Kharkiv Region
  - Research Site, Kirovohrad
  - Research Site, Kyiv
  - Research Site, Liutizh
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Sumy
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
- United Kingdom (7):
  - Research Site, Guildford
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Nottingham
  - Research Site, Taunton
  - Research Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Cheng Y, Zhou Q, Han B, Fan Y, Shan L, Chang J, Sun S, Fang J, Chen Y, Sun J, Wu G, Mann H, Naicker K, Shire N, Mok T, de Castro G Jr. NEPTUNE China cohort: First-line durvalumab plus tremelimumab in Chinese patients with metastatic non-small-cell lung cancer. Lung Cancer. 2023 Apr;178:87-95. doi: 10.1016/j.lungcan.2023.01.013. Epub 2023 Feb 1. PMID 36806898
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419AC00003&attachmentIdentifier=8b9563bd-cf14-4923-8681-fa20813a5b58&fileName=D419AC00003_(Neptune)_Clinical_Study_Protocol_V9.0_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419AC00003&attachmentIdentifier=9e32a3a4-86d6-47b0-b0f2-852ff8a9c707&fileName=D419AC00003_(Neptune)_Statistical_Analysis_Plan_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 192 centers across 29 countries in North America, Latin America, Asia, Europe and Gulf countries randomized adults with epidermal growth factor receptor and anaplastic lymphoma kinase wild-type advanced or metastatic non-small-cell lung cancer (NSCLC) in this study. First participant was enrolled on 03 November 2015 and final data cut-off (DCO) date was 24 June 2019 for Global cohort and 21 September 2020 for China cohort. SoC = standard of care
Pre-assignment Details: 823 participants in Global cohort and 160 participants in China cohort were randomized in 1:1 ratio to receive durvalumab + tremelimumab or SoC chemotherapy. China cohort comprised participants from mainland China (30 from Global cohort and 130 randomized after end of Global cohort recruitment). Thus, 953 unique participants were randomized in the study overall. Participants included in both cohorts for Started, Completed and Reasons for Not Completed are not double-counted for participant flow.
Groups:
- All Participants: Durvalumab + Tremelimumab: Participants received durvalumab 20 milligram per kilogram (mg/kg) and tremelimumab 1 mg/kg intravenous (IV) infusion every 4 weeks (Q4W) in combination for up to 4 doses/cycles. Participants then continued to receive durvalumab 20 mg/kg Q4W, starting on Week 16 until objective disease progression (PD), initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or specific treatment discontinuation criteria were met.
- All Participants: SoC Chemotherapy: Participants received 1 of the following IV infusion treatment combinations on Day 1 of each 21-day cycle for 4 to 6 cycles or until objective PD, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or specific treatment discontinuation criteria were met.
  1. Paclitaxel 200 mg/square meter (m^2) and carboplatin area under the plasma concentration curve (AUC) 5 or 6 mg*minute per milliliter (mg*min/mL).
  2. Gemcitabine 1000 or 1250 mg/m^2 and cisplatin 75 or 80 mg/m^2. Additional dose of gemcitabine 1000 or 1250 mg/m^2 on Day 8 of each cycle (For squamous participants only).
  3. Gemcitabine 1000 or 1250 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL. Additional dose of gemcitabine 1000 or 1250 mg/m^2 on Day 8 of each cycle (For squamous participants only).
  4. Pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2 (For non-squamous participants only; pemetrexed maintenance dose was permitted).
  5. Pemetrexed 500 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL (For non-squamous participants only; pemetrexed maintenance dose was permitted).
Period: Overall Study
Arm/Group | All Participants: Durvalumab + Tremelimumab | All Participants: SoC Chemotherapy
Started (Randomized in overall study) | 474 | 479
Randomized in Global Cohort | 410 | 413
Received Treatment in Global Cohort | 410 | 399
Randomized in China Cohort | 78 | 82
Received Treatment in China Cohort | 77 | 78
Included in Both Cohorts (Global and China) | 14 | 16
Ongoing in Study at DCO for Final Analysis in Global Cohort | 75 | 67
Ongoing in Study at DCO for Final Analysis in China Cohort | 27 | 18
Completed (Ongoing in overall study at DCO for final analysis.) | 99 | 83
Not Completed | 375 | 396
Not completed — Death | 367 | 377
Not completed — Withdrawal by Subject | 8 | 19

BASELINE CHARACTERISTICS:
Population: Global Cohort: The full analysis set (FAS) included all randomized participants prior to the end of global recruitment. Any participants recruited in China, after global recruitment had ended, were not included in the FAS.
  China Cohort: The China FAS included all randomized participants in the China cohort and were used for all China only efficacy analyses.
  Participants included in both cohorts are not double-counted for the baseline characteristics analysis represented by 'All participants'.
Groups:
- All Participants: Durvalumab + Tremelimumab: Participants received durvalumab 20 mg/kg and tremelimumab 1 mg/kg IV infusion Q4W in combination for up to 4 doses/cycles. Participants then continued to receive durvalumab 20 mg/kg Q4W, starting on Week 16 until objective PD, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or specific treatment discontinuation criteria were met.
- All Participants: SoC Chemotherapy: Participants received 1 of the following IV infusion treatment combinations on Day 1 of each 21-day cycle for 4 to 6 cycles or until objective PD, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or specific treatment discontinuation criteria were met.
  1. Paclitaxel 200 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL.
  2. Gemcitabine 1000 or 1250 mg/m^2 and cisplatin 75 or 80 mg/m^2. Additional dose of gemcitabine 1000 or 1250 mg/m^2 on Day 8 of each cycle (For squamous participants only).
  3. Gemcitabine 1000 or 1250 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL. Additional dose of gemcitabine 1000 or 1250 mg/m^2 on Day 8 of each cycle (For squamous participants only).
  4. Pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2 (For non-squamous participants only; pemetrexed maintenance dose was permitted).
  5. Pemetrexed 500 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL (For non-squamous participants only; pemetrexed maintenance dose was permitted).
- Total: Total of all reporting groups
Arm/Group | All Participants: Durvalumab + Tremelimumab | All Participants: SoC Chemotherapy | Total
Number analyzed (Participants) | 474 | 479 | 953
Age, Customized [Count of Participants; unit: Participants] — Population: Baseline data is presented for all participants, as well as separately for the Global and China cohorts.
  Participants
    All participants: <=18 years | 0 | 0 | 0
    All participants: Between 18 and 65 years | 278 | 244 | 522
    All participants: >=65 years | 196 | 235 | 431
    Global cohort: number analyzed (Participants) | 410 | 413 | 823
    Global cohort: <=18 years | 0 | 0 | 0
    Global cohort: Between 18 and 65 years | 233 | 203 | 436
    Global cohort: >=65 years | 177 | 210 | 387
    China cohort: number analyzed (Participants) | 78 | 82 | 160
    China cohort: <=18 years | 0 | 0 | 0
    China cohort: Between 18 and 65 years | 53 | 51 | 104
    China cohort: >=65 years | 25 | 31 | 56
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline data is presented for all participants, as well as separately for the Global and China cohorts.
  Participants
    All participants: Female | 127 | 129 | 256
    All participants: Male | 347 | 350 | 697
    Global cohort: number analyzed (Participants) | 410 | 413 | 823
    Global cohort: Female | 113 | 108 | 221
    Global cohort: Male | 297 | 305 | 602
    China cohort: number analyzed (Participants) | 78 | 82 | 160
    China cohort: Female | 18 | 25 | 43
    China cohort: Male | 60 | 57 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline data is presented for all participants, as well as separately for the Global and China cohorts.
  Participants
    All participants: White | 307 | 289 | 596
    All participants: Black or African American | 3 | 7 | 10
    All participants: Asian | 150 | 165 | 315
    All participants: American Indian or Alaska Native | 10 | 12 | 22
    All participants: Other | 3 | 4 | 7
    All participants: Missing | 1 | 2 | 3
    Global cohort: number analyzed (Participants) | 410 | 413 | 823
    Global cohort: White | 307 | 289 | 596
    Global cohort: Black or African American | 3 | 7 | 10
    Global cohort: Asian | 86 | 99 | 185
    Global cohort: American Indian or Alaska Native | 10 | 12 | 22
    Global cohort: Other | 3 | 4 | 7
    Global cohort: Missing | 1 | 2 | 3
    China cohort: number analyzed (Participants) | 78 | 82 | 160
    China cohort: White | 0 | 0 | 0
    China cohort: Black or African American | 0 | 0 | 0
    China cohort: Asian | 78 | 82 | 160
    China cohort: American Indian or Alaska Native | 0 | 0 | 0
    China cohort: Other | 0 | 0 | 0
    China cohort: Missing | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline data is presented for all participants, as well as separately for the Global and China cohorts.
  Participants
    All participants: Hispanic or Latino | 50 | 48 | 98
    All participants: Not Hispanic or Latino | 423 | 429 | 852
    All participants: Missing | 1 | 2 | 3
    Global cohort: number analyzed (Participants) | 410 | 413 | 823
    Global cohort: Hispanic or Latino | 50 | 48 | 98
    Global cohort: Not Hispanic or Latino | 359 | 363 | 722
    Global cohort: Missing | 1 | 2 | 3
    China cohort: number analyzed (Participants) | 78 | 82 | 160
    China cohort: Hispanic or Latino | 0 | 0 | 0
    China cohort: Not Hispanic or Latino | 78 | 82 | 160
    China cohort: Missing | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS); Global Cohort: Blood Tumor Mutational Burden (bTMB) ≥20 Mutations Per Megabase (Mut/Mb) Analysis Set
Description: The OS was defined as the time from the date of randomization until death due to any cause (ie, date of death or censoring - date of randomization + 1). Any participant not known to have died at the time of analysis was censored based on the last recorded date on which the participant was known to be alive. Median OS was calculated using the Kaplan-Meier technique.
Time Frame: From baseline (Day 1, Week 0) until death due to any cause, assessed up to the Global cohort DCO date (a maximum of approximately 44 months).
Population: The bTMB ≥20 mut/Mb analysis set included the subset of participants in the FAS whose blood TMB status was ≥20 mut/Mb at baseline as defined by the GuardantOMNI CDx assay. Only participants randomized in Global cohort were analyzed as bTMB and tissue tumor mutational burden (tTMB) testing was not performed in China cohort.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Global: Durvalumab + Tremelimumab: Participants received durvalumab 20 mg/kg and tremelimumab 1 mg/kg IV infusion Q4W in combination for up to 4 doses/cycles. Participants then continued to receive durvalumab 20 mg/kg Q4W, starting on Week 16 until objective PD, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or specific treatment discontinuation criteria were met.
- Global: SoC Chemotherapy: Participants received 1 of the following IV infusion treatment combinations on Day 1 of each 21-day cycle for 4 to 6 cycles or until objective PD, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or specific treatment discontinuation criteria were met.
  1. Paclitaxel 200 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL.
  2. Gemcitabine 1000 or 1250 mg/m^2 and cisplatin 75 or 80 mg/m^2. Additional dose of gemcitabine 1000 or 1250 mg/m^2 on Day 8 of each cycle (For squamous participants only).
  3. Gemcitabine 1000 or 1250 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL. Additional dose of gemcitabine 1000 or 1250 mg/m^2 on Day 8 of each cycle (For squamous participants only).
  4. Pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2 (For non-squamous participants only; pemetrexed maintenance dose was permitted).
  5. Pemetrexed 500 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL (For non-squamous participants only; pemetrexed maintenance dose was permitted).
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy
Number analyzed (Participants) | 69 | 60
months | 11.7 [8.6 to 15.2] | 9.1 [7.8 to 12.6]
Statistical Analysis 1: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; Global: Durvalumab + Tremelimumab versus (Vs) Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Superiority; p = 0.0808, Log Rank — The 2-sided p-value was calculated using an unstratified log-rank test; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.485 to 1.045] — The HR and confidence interval (CI) were calculated using an unstratified Cox proportional hazards model, with ties handled by the Efron approach

2. Primary Outcome: OS; China Cohort: China Programmed Cell Death Ligand 1 (PD-L1) Negative NSCLC Analysis Set
Description: as for outcome 1
Time Frame: From baseline (Day 1, Week 0) until death due to any cause, assessed up to the China cohort DCO date (a maximum of approximately 44 months).
Population: The China PD-L1-negative population analysis set included the subset of participants in the China FAS whose PD-L1 status was PD-L1-negative at baseline as defined by the Ventana SP263 PD-L1 assay (ie, <1% PD-L1-membrane expression in tumoral tissue). Only participants randomized in China cohort were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- China: Durvalumab + Tremelimumab: Participants received durvalumab 20 mg/kg and tremelimumab 1 mg/kg IV infusion Q4W in combination for up to 4 doses/cycles. Participants then continued to receive durvalumab 20 mg/kg Q4W, starting on Week 16 until objective PD, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or specific treatment discontinuation criteria were met.
- China: SoC Chemotherapy: Participants received 1 of the following IV infusion treatment combinations on Day 1 of each 21-day cycle for 4 to 6 cycles or until objective PD, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or specific treatment discontinuation criteria were met.
  1. Paclitaxel 200 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL.
  2. Gemcitabine 1000 or 1250 mg/m^2 and cisplatin 75 or 80 mg/m^2. Additional dose of gemcitabine 1000 or 1250 mg/m^2 on Day 8 of each cycle (For squamous participants only).
  3. Gemcitabine 1000 or 1250 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL. Additional dose of gemcitabine 1000 or 1250 mg/m^2 on Day 8 of each cycle (For squamous participants only).
  4. Pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2 (For non-squamous participants only; pemetrexed maintenance dose was permitted).
  5. Pemetrexed 500 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL (For non-squamous participants only; pemetrexed maintenance dose was permitted).
Arm/Group | China: Durvalumab + Tremelimumab | China: SoC Chemotherapy
Number analyzed (Participants) | 26 | 29
months | 15.0 [10.5 to 27.4] | 11.7 [8.6 to 20.5]
Statistical Analysis 1: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Other — The study was not designed or powered to show statistical significance for efficacy endpoints in the China cohort, so all statistical analyses for the China cohort were considered exploratory; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.322 to 1.109] — The HR and CI were calculated using a stratified Cox proportional hazards model, adjusting for histology (squamous Vs non-squamous), with ties handled by the Efron approach

3. Secondary Outcome: OS; Global Cohort: bTMB ≥16 Mut/Mb, bTMB ≥12 Mut/Mb, PD-L1-Negative NSCLC, bTMB <20 Mut/Mb, bTMB Non-Evaluable Population, tTMB ≥14 Mut/Mb, tTMB ≥12 Mut/Mb, tTMB ≥10 Mut/Mb, and tTMB ≥8 Mut/Mb Analysis Sets
Description: OS was defined as time from date of randomization until death due to any cause (ie, date of death or censoring - date of randomization + 1). Any participant not known to have died at time of analysis was censored based on last recorded date on which participant was known to be alive.
  bTMB ≥16 mut/Mb, bTMB ≥12 mut/Mb and bTMB <20 mut/Mb analysis sets included the subset of participants in FAS whose bTMB status was ≥16 mut/Mb, ≥12 mut/Mb and <20 mut/Mb, respectively at baseline as defined by the GuardantOMNI CDx assay.
  PD-L1-negative analysis set included the subset of participants in FAS whose PD-L1 status was PD-L1-negative at baseline as defined by the Ventana SP263 PD-L1 Assay (ie, <1% PD-L1-membrane expression in tumoral tissue).
  bTMB non-evaluable analysis set included the subset of participants in FAS whose bTMB status at baseline could not be determined by the GuardantOMNI CDx assay or whose sample was not available.
  tTMB analysis sets are defined same as the bTMB analysis sets.
Time Frame: as for outcome 1
Population: Participants included in bTMB ≥16 mut/Mb, bTMB ≥12 mut/Mb, PD-L1-Negative NSCLC, bTMB <20 mut/Mb, bTMB non-evaluable population, tTMB ≥14 mut/Mb, tTMB ≥12 mut/Mb, tTMB ≥10 mut/Mb, and tTMB ≥8 mut/Mb analysis sets are reported in this outcome measure. Only participants randomized in Global cohort were analyzed as bTMB and tTMB testing was not performed in China cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy
Number analyzed (Participants) | 410 | 413
months
  bTMB ≥16 mut/Mb analysis set: number analyzed (Participants) | 93 | 89
  bTMB ≥16 mut/Mb analysis set | 12.1 [8.6 to 15.0] | 11.9 [8.5 to 15.9]
  bTMB ≥12 mut/Mb analysis set: number analyzed (Participants) | 143 | 138
  bTMB ≥12 mut/Mb analysis set | 10.9 [8.6 to 12.6] | 10.3 [8.3 to 12.9]
  PD-L1 negative analysis set: number analyzed (Participants) | 91 | 104
  PD-L1 negative analysis set | 11.1 [8.1 to 14.7] | 12.5 [9.9 to 16.2]
  bTMB <20 mut/Mb analysis set: number analyzed (Participants) | 197 | 186
  bTMB <20 mut/Mb analysis set | 9.9 [7.7 to 12.8] | 11.5 [8.8 to 13.7]
  bTMB non-evaluable analysis set: number analyzed (Participants) | 111 | 123
  bTMB non-evaluable analysis set | 9.3 [7.2 to 15.5] | 10.4 [9.4 to 13.8]
  tTMB ≥14 mut/Mb analysis set: number analyzed (Participants) | 31 | 38
  tTMB ≥14 mut/Mb analysis set | 17.5 [9.8 to NA] — Upper limit was not reached. | 10.6 [7.0 to 20.9]
  tTMB ≥12 mut/Mb analysis set: number analyzed (Participants) | 54 | 55
  tTMB ≥12 mut/Mb analysis set | 11.1 [7.0 to 17.5] | 13.9 [9.0 to 17.9]
  tTMB ≥10 mut/Mb analysis set: number analyzed (Participants) | 77 | 80
  tTMB ≥10 mut/Mb analysis set | 11.1 [7.2 to 15.7] | 10.6 [9.0 to 15.7]
  tTMB ≥8 mut/Mb analysis set: number analyzed (Participants) | 90 | 97
  tTMB ≥8 mut/Mb analysis set | 11.0 [7.8 to 15.7] | 10.2 [8.0 to 13.5]
Statistical Analysis 1: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥16 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.629 to 1.201] — The HR and CI were calculated using an unstratified Cox proportional hazards model, with ties handled by the Efron approach
Statistical Analysis 2: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥12 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.726 to 1.213] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; PD-L1 negative analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Superiority; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.786 to 1.464] — The HR and CI were calculated using a stratified Cox proportional hazards model, adjusting for smoking status (never smoker Vs ever smoker) and histology (squamous Vs non-squamous), with ties handled by the Efron approach
Statistical Analysis 4: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB <20 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Superiority; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.835 to 1.302] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB non-evaluable analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Superiority; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.758 to 1.353] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; tTMB ≥14 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.309 to 1.008] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; tTMB ≥12 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.560 to 1.350] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; tTMB ≥10 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.614 to 1.251] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; tTMB ≥8 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.564 to 1.080] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: OS; Global and China Cohorts: FAS, PD-L1 Tumor Cell (TC) ≥25%, and PD-L1 TC ≥50% Analysis Sets
Description: The OS was defined as time from date of randomization until death due to any cause (ie, date of death or censoring - date of randomization + 1). Any participant not known to have died at the time of analysis was censored based on last recorded date on which participant was known to be alive.
  Global Cohort: The FAS included all randomized participants prior to the end of global recruitment. Any participants recruited in China, after global recruitment had ended, were not included in the FAS.
  China Cohort: The China FAS included all randomized participants in the China cohort and were used for all China only efficacy analyses.
  PD-L1 TC ≥25% and PD-L1 TC ≥50% analysis sets included the subset of participants in the FAS whose PD-L1 status was TC ≥25% and TC ≥50% membrane expression in tumoral tissue, respectively at baseline as defined by the Ventana SP263 PD-L1 Assay.
Time Frame: From baseline (Day 1, Week 0) until death due to any cause, assessed up to the Global or China cohort DCO dates, as applicable (a maximum of approximately 44 months) for each cohort.
Population: Participants included in FAS, PD-L1 TC ≥25%, and PD-L1 TC ≥50% analysis sets are reported in this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy | China: Durvalumab + Tremelimumab | China: SoC Chemotherapy
Number analyzed (Participants) | 410 | 413 | 78 | 82
months
  FAS | 10.9 [9.3 to 12.6] | 12.1 [10.3 to 13.5] | 20.0 [15.0 to 28.7] | 14.1 [9.5 to 19.4]
  PD-L1 TC ≥25% analysis set: number analyzed (Participants) | 165 | 164 | 31 | 32
  PD-L1 TC ≥25% analysis set | 12.2 [9.7 to 15.2] | 10.4 [8.6 to 12.2] | 36.6 [15.5 to NA] — Upper limit was not reached. | 15.8 [9.0 to 26.9]
  PD-L1 TC ≥50% analysis set: number analyzed (Participants) | 115 | 116 | 25 | 28
  PD-L1 TC ≥50% analysis set | 14.1 [10.0 to 19.3] | 10.5 [8.7 to 12.6] | 36.6 [16.9 to NA] — Upper limit was not reached. | 15.8 [9.0 to 26.9]
Statistical Analysis 1: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; FAS: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Superiority; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.871 to 1.186] — The HR and CI were calculated using a stratified Cox proportional hazards model, adjusting for PD-L1 status (≥25% Vs <25%), smoking status (never smoker Vs ever smoker) and histology (squamous Vs non-squamous), with ties handled by Efron approach
Statistical Analysis 2: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; FAS: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.480 to 1.018] — The HR and CI were calculated using a stratified Cox proportional hazards model, adjusting for PD-L1 status (>= 25% Vs < 25 and histology (squamous Vs non-squamous), with ties handled by the Efron approach
Statistical Analysis 3: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; PD-L1 TC ≥25% analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.654 to 1.078] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 4: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; PD-L1 TC ≥ 25% analysis set: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.289 to 1.065] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; PD-L1 TC ≥50% analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.587 to 1.081] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 6: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; PD-L1 TC ≥50% analysis set: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer OS than SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.222 to 0.955] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Progression-Free Survival (PFS); Global Cohort: bTMB ≥20 Mut/Mb, bTMB ≥16 Mut/Mb, bTMB ≥12 Mut/Mb, tTMB ≥14 Mut/Mb, tTMB ≥12 Mut/Mb, tTMB ≥10 Mut/Mb, and tTMB ≥8 Mut/Mb Analysis Sets
Description: The PFS (per Response Evaluation Criteria in Solid Tumors, version 1.1 [RECIST 1.1] using Investigator assessments) was defined as the time from the date of randomization until the date of objective PD or death (by any cause in the absence of progression) regardless of whether the participant withdrew from randomized therapy or received another anticancer therapy prior to progression (ie, date of PFS event or censoring - date of randomization + 1).
  bTMB ≥20 mut/Mb, bTMB ≥16 mut/Mb and bTMB ≥12 mut/Mb analysis sets included the subset of participants in FAS whose bTMB status was ≥20 mut/Mb, ≥16 mut/Mb and ≥12 mut/Mb, respectively at baseline as defined by the GuardantOMNI CDx assay.
  tTMB ≥14 mut/Mb, tTMB ≥12 mut/Mb, tTMB ≥10 mut/Mb and tTMB ≥8 mut/Mb analysis sets included the subset of participants in FAS whose tTMB status was ≥14 mut/Mb, ≥12 mut/Mb, ≥10 mut/Mb and ≥8 mut/Mb, respectively at baseline as defined by the GuardantOMNI CDx assay.
Time Frame: Tumour scans performed at baseline and every 6 weeks up to 48 weeks relative to date of randomization, then every 8 weeks thereafter until confirmed PD/death. Up to Global cohort DCO date (approximately 44 months).
Population: Participants included in bTMB ≥20 mut/Mb, bTMB ≥16 mut/Mb, bTMB ≥12 mut/Mb, tTMB ≥14 mut/Mb, tTMB ≥12 mut/Mb, tTMB ≥10 mut/Mb, and tTMB ≥8 mut/Mb analysis sets are reported in this outcome measure. Only participants randomized in Global cohort were analyzed as bTMB and tTMB testing was not performed in China cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy
Number analyzed (Participants) | 410 | 413
months
  bTMB ≥20 mut/Mb analysis set: number analyzed (Participants) | 69 | 60
  bTMB ≥20 mut/Mb analysis set | 4.2 [2.7 to 5.6] | 5.1 [4.2 to 5.6]
  bTMB ≥16 mut/Mb analysis set: number analyzed (Participants) | 93 | 89
  bTMB ≥16 mut/Mb analysis set | 4.2 [2.8 to 5.5] | 5.5 [4.4 to 5.8]
  bTMB ≥12 mut/Mb analysis set: number analyzed (Participants) | 143 | 138
  bTMB ≥12 mut/Mb analysis set | 3.9 [2.8 to 4.8] | 5.1 [4.4 to 5.6]
  tTMB ≥14 mut/Mb analysis set: number analyzed (Participants) | 31 | 38
  tTMB ≥14 mut/Mb analysis set | 8.7 [5.2 to 22.3] | 5.8 [4.4 to 7.9]
  tTMB ≥12 mut/Mb analysis set: number analyzed (Participants) | 54 | 55
  tTMB ≥12 mut/Mb analysis set | 5.2 [3.8 to 6.9] | 5.8 [4.2 to 6.6]
  tTMB ≥10 mut/Mb analysis set: number analyzed (Participants) | 77 | 80
  tTMB ≥10 mut/Mb analysis set | 4.3 [2.8 to 5.5] | 5.1 [4.2 to 5.8]
  tTMB ≥8 mut/Mb analysis set: number analyzed (Participants) | 90 | 97
  tTMB ≥8 mut/Mb analysis set | 4.4 [2.9 to 5.5] | 5.0 [4.2 to 5.6]
Statistical Analysis 1: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥20 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.514 to 1.146] — The HR and CI interval were calculated using an unstratified Cox proportional hazards model, with ties handled by the Efron approach
Statistical Analysis 2: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥16 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.623 to 1.189] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥12 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.714 to 1.193] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; tTMB ≥14 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.258 to 0.818] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; tTMB ≥12 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.524 to 1.228] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; tTMB ≥10 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.585 to 1.177] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; tTMB ≥8 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.534 to 1.017] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: PFS; Global and China Cohorts: PD-L1-Negative NSCLC, FAS, PD-L1 TC ≥25%, and PD-L1 TC ≥50% Analysis Sets
Description: PFS (per RECIST 1.1 using Investigator assessments) was defined as time from date of randomization until date of objective PD or death regardless of whether participant withdrew from randomized therapy or received another anticancer therapy prior to progression (ie, date of PFS event or censoring - date of randomization + 1).
  PD-L1-negative analysis set included subset of participants in FAS whose PD-L1 status was PD-L1-negative at baseline as defined by Ventana SP263 PD-L1 Assay (ie, <1% PD-L1-membrane expression in tumoral tissue).
  Global Cohort: FAS included all randomized participants prior to end of global recruitment.
  China Cohort: China FAS included all randomized participants in China cohort and were used for all China only efficacy analyses.
  PD-L1 TC ≥25% and PD-L1 TC ≥50% analysis sets included subset of participants in FAS whose PD-L1 status was TC ≥25% and TC ≥50% membrane expression in tumoral tissue, respectively at baseline as defined by the Ventana SP263 PD-L1 Assay.
Time Frame: Tumour scans performed at baseline and every 6 weeks up to 48 weeks relative to date of randomization, then every 8 weeks thereafter until confirmed PD/death. Up to Global or China cohort DCO dates, as applicable (approximately 44 months) for each cohort.
Population: Participants included in PD-L1-negative NSCLC, FAS, PD-L1 TC ≥25%, and PD-L1 TC ≥50% analysis sets are reported in this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy | China: Durvalumab + Tremelimumab | China: SoC Chemotherapy
Number analyzed (Participants) | 410 | 413 | 78 | 82
months
  PD-L1-negative NSCLC analysis set: number analyzed (Participants) | 91 | 104 | 26 | 29
  PD-L1-negative NSCLC analysis set | 4.1 [2.8 to 5.2] | 5.6 [4.6 to 6.0] | 5.1 [2.8 to 7.2] | 6.0 [4.0 to 7.5]
  FAS | 4.0 [2.9 to 4.2] | 5.6 [5.3 to 5.7] | 4.2 [2.8 to 7.2] | 6.0 [5.5 to 7.5]
  PD-L1 TC ≥25% analysis set: number analyzed (Participants) | 165 | 164 | 31 | 32
  PD-L1 TC ≥25% analysis set | 4.2 [3.2 to 5.7] | 5.4 [4.4 to 5.6] | 6.8 [4.1 to 8.4] | 5.7 [4.2 to 8.5]
  PD-L1 TC ≥50% analysis set: number analyzed (Participants) | 115 | 116 | 25 | 28
  PD-L1 TC ≥50% analysis set | 4.6 [3.1 to 6.0] | 5.4 [4.3 to 5.6] | 6.8 [4.2 to 20.2] | 5.7 [4.2 to 8.5]
Statistical Analysis 1: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; PD-L1-negative analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Superiority; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.810 to 1.517] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 2: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; PD-L1-negative analysis set: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.592 to 2.141] — The HR and CI interval were calculated using an stratified Cox proportional hazards model, adjusting histology (squamous Vs non-squamous), with ties handled by the Efron approach
Statistical Analysis 3: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; FAS: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Superiority; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.924 to 1.253] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; FAS: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.655 to 1.362] — The HR and CI were calculated using a stratified Cox proportional hazards model, adjusting for PD-L1 status (≥ 25% Vs < 25%) and histology (squamous Vs non-squamous), with ties handled by the Efron approach
Statistical Analysis 5: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; PD-L1 TC ≥25% analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.621 to 1.024] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 6: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; PD-L1 TC ≥ 25% analysis set: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.389 to 1.317] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; PD-L1 TC ≥50% analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.542 to 1.010] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 8: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; PD-L1 TC ≥50% analysis set: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer PFS than SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.335 to 1.251] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Objective Response Rate (ORR); Global Cohort: bTMB ≥20 Mut/Mb, bTMB ≥16 Mut/Mb, bTMB ≥12 Mut/Mb, tTMB ≥14 Mut/Mb, tTMB ≥12 Mut/Mb, tTMB ≥10 Mut/Mb, and tTMB ≥8 Mut/Mb Analysis Sets
Description: The ORR (per RECIST 1.1 using Investigator assessments) was defined as the percentage of participants with at least 1 visit response of complete response (CR) or partial response (PR) prior to PD.
  bTMB ≥20 mut/Mb, bTMB ≥16 mut/Mb and bTMB ≥12 mut/Mb analysis sets included the subset of participants in FAS whose bTMB status was ≥20 mut/Mb, ≥16 mut/Mb and ≥12 mut/Mb, respectively at baseline as defined by the GuardantOMNI CDx assay.
  tTMB ≥14 mut/Mb, tTMB ≥12 mut/Mb, tTMB ≥10 mut/Mb and tTMB ≥8 mut/Mb analysis sets included the subset of participants in FAS whose tTMB status was ≥14 mut/Mb, ≥12 mut/Mb, ≥10 mut/Mb and ≥8 mut/Mb, respectively at baseline as defined by the GuardantOMNI CDx assay.
Time Frame: as for outcome 5
Population: Participants included in bTMB ≥20 mut/Mb, bTMB ≥16 mut/Mb, bTMB ≥12 mut/Mb, tTMB ≥14 mut/Mb, tTMB ≥12 mut/Mb, tTMB ≥10 mut/Mb, and tTMB ≥8 mut/Mb analysis sets with measurable disease are reported in this outcome measure. Only participants randomized in Global cohort were analyzed as bTMB and tTMB testing was not performed in China cohort.
Measure: Number; unit: percentage of participants
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy
Number analyzed (Participants) | 410 | 413
percentage of participants
  bTMB ≥20 mut/Mb analysis set: number analyzed (Participants) | 69 | 60
  bTMB ≥20 mut/Mb analysis set | 27.5 | 43.3
  bTMB ≥16 mut/Mb analysis set: number analyzed (Participants) | 93 | 89
  bTMB ≥16 mut/Mb analysis set | 31.2 | 46.1
  bTMB ≥12 mut/Mb analysis set: number analyzed (Participants) | 143 | 138
  bTMB ≥12 mut/Mb analysis set | 28.7 | 42.0
  tTMB ≥14 mut/Mb analysis set: number analyzed (Participants) | 31 | 38
  tTMB ≥14 mut/Mb analysis set | 61.3 | 44.7
  tTMB ≥12 mut/Mb analysis set: number analyzed (Participants) | 54 | 55
  tTMB ≥12 mut/Mb analysis set | 42.6 | 41.8
  tTMB ≥10 mut/Mb analysis set: number analyzed (Participants) | 77 | 80
  tTMB ≥10 mut/Mb analysis set | 37.7 | 42.5
  tTMB ≥8 mut/Mb analysis set: number analyzed (Participants) | 90 | 97
  tTMB ≥8 mut/Mb analysis set | 36.7 | 41.2
Statistical Analysis 1: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥20 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Superiority; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.236 to 1.030]
Statistical Analysis 2: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥16 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Superiority; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.288 to 0.968]
Statistical Analysis 3: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥12 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Superiority; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.336 to 0.908]
Statistical Analysis 4: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; tTMB ≥14 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Superiority; Odds Ratio (OR) = 1.96, 95% CI 2-sided [0.752 to 5.234]
Statistical Analysis 5: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; tTMB ≥12 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Superiority; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.482 to 2.214]
Statistical Analysis 6: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; tTMB ≥10 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Superiority; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.430 to 1.548]
Statistical Analysis 7: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; tTMB ≥8 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Superiority; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.456 to 1.486]

8. Secondary Outcome: ORR; Global and China Cohorts: PD-L1-Negative NSCLC, FAS, PD-L1 TC ≥25%, and PD-L1 TC ≥50% Analysis Sets
Description: The ORR (per RECIST 1.1 using Investigator assessments) was defined as the percentage of participants with at least 1 visit response of CR or PR prior to PD.
  PD-L1-negative analysis set included the subset of participants in FAS whose PD-L1 status was PD-L1-negative at baseline as defined by the Ventana SP263 PD-L1 Assay (ie, <1% PD-L1-membrane expression in tumoral tissue).
  Global Cohort: The FAS included all randomized participants prior to the end of global recruitment.
  China Cohort: The China FAS included all randomized participants in the China cohort and were used for all China only efficacy analyses.
  PD-L1 TC ≥25% and PD-L1 TC ≥50% analysis sets included the subset of participants in the FAS whose PD-L1 status was TC ≥25% and TC ≥50% membrane expression in tumoral tissue, respectively at baseline as defined by the Ventana SP263 PD-L1 Assay.
Time Frame: as for outcome 6
Population: Participants included in PD-L1-negative NSCLC, FAS, PD-L1 TC ≥25%, and PD-L1 TC ≥50% analysis sets with measurable disease are reported in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy | China: Durvalumab + Tremelimumab | China: SoC Chemotherapy
Number analyzed (Participants) | 410 | 413 | 78 | 82
percentage of participants
  PD-L1-negative NSCLC analysis set: number analyzed (Participants) | 91 | 103 | 26 | 29
  PD-L1-negative NSCLC analysis set | 23.1 | 38.8 | 23.1 | 41.4
  FAS: number analyzed (Participants) | 410 | 412 | 78 | 82
  FAS | 25.9 | 41.7 | 35.9 | 39.0
  PD-L1 TC ≥25% analysis set: number analyzed (Participants) | 165 | 164 | 31 | 32
  PD-L1 TC ≥25% analysis set | 35.2 | 43.9 | 54.8 | 40.6
  PD-L1 TC ≥50% analysis set: number analyzed (Participants) | 115 | 116 | 25 | 28
  PD-L1 TC ≥50% analysis set | 37.4 | 44.0 | 60.0 | 46.4
Statistical Analysis 1: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; PD-L1-negative analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Superiority; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.245 to 0.869] — The analysis was performed using logistic regression, adjusting for smoking status (never smoker Vs ever smoker) and histology (squamous Vs non-squamous), with 95% CI calculated by profile likelihood
Statistical Analysis 2: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; PD-L1-negative analysis set: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Binomial exact test; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.124 to 1.337]
Statistical Analysis 3: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; FAS: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Superiority; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.356 to 0.647] — The analysis was performed using logistic regression adjusting for PD-L1 status (≥25% Vs <25%), smoking status (never smoker Vs ever smoker) and histology (squamous Vs non-squamous), with 95% CI calculated by profile likelihood
Statistical Analysis 4: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; FAS: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.450 to 1.660] — The analysis was performed using logistic regression, adjusting for PD-L1 status (>= 25% Vs < 25%), smoking status (never smoker Va ever smoker) and histology (squamous Vs non-squamous), with 95% CI calculated by profile likelihood
Statistical Analysis 5: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; PD-L1 TC ≥25% analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Superiority; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.443 to 1.079] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; PD-L1 TC ≥ 25% analysis set: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.658 to 4.919] — [estimate comment as in outcome 8, analysis 4]
Statistical Analysis 7: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; PD-L1 TC ≥50% analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Superiority; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.449 to 1.291] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 8: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; PD-L1 TC ≥50% analysis set: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy An odds ratio >1 favors Durvalumab + Tremelimumab combination therapy over SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.585 to 5.270] — [estimate comment as in outcome 8, analysis 4]

9. Secondary Outcome: Duration of Response (DoR); Global Cohort: bTMB ≥20 Mut/Mb, bTMB ≥16 Mut/Mb, and bTMB ≥12 Mut/Mb Analysis Sets
Description: DoR (per RECIST 1.1 using Investigator assessments) was defined as the time from the date of first documented response (CR or PR) until the first date of documented progression or death in the absence of PD (ie, date of PFS event or censoring - date of first response + 1).
  bTMB ≥20 mut/Mb, bTMB ≥16 mut/Mb and bTMB ≥12 mut/Mb analysis sets included the subset of participants in FAS whose bTMB status was ≥20 mut/Mb, ≥16 mut/Mb and ≥12 mut/Mb, respectively at baseline as defined by the GuardantOMNI CDx assay.
Time Frame: as for outcome 5
Population: Participants included in bTMB ≥20 mut/Mb, bTMB ≥16 mut/Mb, and bTMB ≥12 mut/Mb analysis sets are reported in this outcome measure. Only participants with objective response and randomized in Global cohort were analyzed as bTMB and tTMB testing was not performed in China cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy
Number analyzed (Participants) | 106 | 172
months
  bTMB ≥20 mut/Mb analysis set: number analyzed (Participants) | 19 | 26
  bTMB ≥20 mut/Mb analysis set | 11.6 [6.7 to 21.5] | 4.2 [3.0 to 6.9]
  bTMB ≥16 mut/Mb analysis set: number analyzed (Participants) | 29 | 41
  bTMB ≥16 mut/Mb analysis set | 10.6 [4.2 to 21.5] | 4.3 [3.0 to 5.9]
  bTMB ≥12 mut/Mb analysis set: number analyzed (Participants) | 41 | 58
  bTMB ≥12 mut/Mb analysis set | 11.5 [6.7 to 18.8] | 4.3 [3.0 to 5.6]
Statistical Analysis 1: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥20 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer DoR than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.25, 95% CI 2-sided [0.113 to 0.532] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥16 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer DoR than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.196 to 0.639] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥12 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer DoR than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.38, 95% CI 2-sided [0.233 to 0.611] — [estimate comment as in outcome 3, analysis 1]

10. Secondary Outcome: DoR; Global and China Cohorts: PD-L1-Negative NSCLC and FAS Analysis Sets
Description: DoR (per RECIST 1.1 using Investigator assessments) was defined as the time from the date of first documented response (CR or PR) until the first date of documented progression or death in the absence of PD (ie, date of PFS event or censoring - date of first response + 1).
  PD-L1-negative analysis set included the subset of participants in FAS whose PD-L1 status was PD-L1-negative at baseline as defined by the Ventana SP263 PD-L1 Assay (ie, <1% PD-L1-membrane expression in tumoral tissue).
  Global Cohort: The FAS included all randomized participants prior to the end of global recruitment.
  China Cohort: The China FAS included all randomized participants in the China cohort and were used for all China only efficacy analyses.
Time Frame: as for outcome 6
Population: Participants included in PD-L1-negative NSCLC and FAS analysis sets are reported in this outcome measure. Only participants with objective response were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy | China: Durvalumab + Tremelimumab | China: SoC Chemotherapy
Number analyzed (Participants) | 106 | 172 | 28 | 32
months
  PD-L1-negative NSCLC analysis set: number analyzed (Participants) | 21 | 40 | 6 | 12
  PD-L1-negative NSCLC analysis set | 10.2 [2.8 to 18.8] | 4.9 [4.2 to 6.1] | 10.5 [1.4 to NA] — Upper limit was not reached. | 6.1 [3.0 to 11.7]
  FAS | 11.1 [6.9 to 15.2] | 4.9 [4.2 to 5.6] | 12.9 [5.4 to 33.6] | 6.1 [4.4 to 7.2]
Statistical Analysis 1: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; PD-L1-negative analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer DoR than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.199 to 0.787] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 2: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; PD-L1-negative analysis set: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer DoR than SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.183 to 2.860] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; FAS: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer DoR than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.324 to 0.588] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; FAS: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab combination therapy to be associated with a longer DoR than SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.193 to 0.761] — The HR and CI were calculated using a stratified Cox proportional hazards model, adjusting for PD-L1 status (>= 25% Vs < 25%) and histology (squamous Vs non-squamous), with ties handled by the Efron approach

11. Secondary Outcome: Alive and Progression-Free at 12 Months (APF12); Global Cohort: bTMB ≥20 Mut/Mb, bTMB ≥16 Mut/Mb, and bTMB ≥12 Mut/Mb Analysis Sets
Description: The APF12 was defined as the percentage of participants who were alive and progression free at 12 months from randomization (ie, PFS rate at 12 months).
  bTMB ≥20 mut/Mb, bTMB ≥16 mut/Mb and bTMB ≥12 mut/Mb analysis sets included the subset of participants in FAS whose bTMB status was ≥20 mut/Mb, ≥16 mut/Mb and ≥12 mut/Mb, respectively at baseline as defined by the GuardantOMNI CDx assay.
Time Frame: Tumour scans performed at baseline then every 6 weeks up to 12 months.
Population: Participants included in bTMB ≥20 mut/Mb, bTMB ≥16 mut/Mb, and bTMB ≥12 mut/Mb analysis sets are reported in this outcome measure. Only participants randomized in Global cohort were analyzed as bTMB and tTMB testing was not performed in China cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy
Number analyzed (Participants) | 143 | 138
percentage of participants
  bTMB ≥20 mut/Mb analysis set: number analyzed (Participants) | 69 | 60
  bTMB ≥20 mut/Mb analysis set | 25.6 [15.7 to 36.6] | 7.0 [1.9 to 16.8]
  bTMB ≥16 mut/Mb analysis set: number analyzed (Participants) | 93 | 89
  bTMB ≥16 mut/Mb analysis set | 22.0 [14.1 to 31.1] | 12.3 [6.1 to 20.8]
  bTMB ≥12 mut/Mb analysis set | 21.6 [15.2 to 28.9] | 13.8 [8.3 to 20.6]

12. Secondary Outcome: APF12; Global and China Cohorts: PD-L1-Negative NSCLC and FAS Analysis Sets
Description: The APF12 was defined as the percentage of patients who were alive and progression free at 12 months from randomization (ie, PFS rate at 12 months).
  PD-L1-negative analysis set included the subset of participants in FAS whose PD-L1 status was PD-L1-negative at baseline as defined by the Ventana SP263 PD-L1 Assay (ie, <1% PD-L1-membrane expression in tumoral tissue).
  Global Cohort: The FAS included all randomized participants prior to the end of global recruitment.
  China Cohort: The China FAS included all randomized participants in the China cohort and were used for all China only efficacy analyses.
Time Frame: Tumour scans performed at baseline then every 6 weeks up to 12 months.
Population: Participants included in PD-L1-negative NSCLC and FAS analysis sets are reported in this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy | China: Durvalumab + Tremelimumab | China: SoC Chemotherapy
Number analyzed (Participants) | 410 | 413 | 78 | 82
percentage of participants
  PD-L1-negative NSCLC analysis set: number analyzed (Participants) | 91 | 104 | 26 | 29
  PD-L1-negative NSCLC analysis set | 18.2 [10.9 to 26.9] | 12.1 [6.3 to 19.9] | 15.6 [4.0 to 34.4] | 11.3 [2.3 to 28.5]
  FAS | 20.2 [16.4 to 24.3] | 14.9 [11.4 to 18.9] | 23.9 [14.8 to 34.2] | 16.6 [8.5 to 27.0]

13. Secondary Outcome: Time From Randomization to Second Progression or Death (PFS2); Global Cohort: bTMB ≥20 Mut/Mb, bTMB ≥16 Mut/Mb, and bTMB ≥12 Mut/Mb Analysis Sets
Description: The PFS2 was defined as the time from the date of randomization to the earliest of the progression events subsequent to that used for the primary variable PFS, or death (ie, date of PFS2 event or censoring - date of randomization + 1).
  bTMB ≥20 mut/Mb, bTMB ≥16 mut/Mb and bTMB ≥12 mut/Mb analysis sets included the subset of participants in FAS whose bTMB status was ≥20 mut/Mb, ≥16 mut/Mb and ≥12 mut/Mb, respectively at baseline as defined by the GuardantOMNI CDx assay.
Time Frame: as for outcome 5
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy
Number analyzed (Participants) | 143 | 138
months
  bTMB ≥20 mut/Mb analysis set: number analyzed (Participants) | 69 | 60
  bTMB ≥20 mut/Mb analysis set | 10.6 [8.5 to 14.4] | 8.6 [7.3 to 12.6]
  bTMB ≥16 mut/Mb analysis set: number analyzed (Participants) | 93 | 89
  bTMB ≥16 mut/Mb analysis set | 10.9 [8.5 to 14.1] | 10.5 [8.0 to 13.2]
  bTMB ≥12 mut/Mb analysis set | 9.9 [8.2 to 11.7] | 9.0 [7.8 to 10.8]
Statistical Analysis 1: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥20 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab to be associated with a longer time to second progression than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.494 to 1.058] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥16 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab to be associated with a longer time to second progression than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.607 to 1.151] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; bTMB ≥12 mut/Mb analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab to be associated with a longer time to second progression than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.689 to 1.146] — [estimate comment as in outcome 3, analysis 1]

14. Secondary Outcome: PFS2; Global and China Cohorts: PD-L1-Negative NSCLC and FAS Analysis Sets
Description: The PFS2 was defined as the time from the date of randomization to the earliest of the progression events subsequent to that used for the primary variable PFS, or death (ie, date of PFS2 event or censoring - date of randomization + 1).
  PD-L1-negative analysis set included the subset of participants in FAS whose PD-L1 status was PD-L1-negative at baseline as defined by the Ventana SP263 PD-L1 Assay (ie, <1% PD-L1-membrane expression in tumoral tissue).
  Global Cohort: The FAS included all randomized participants prior to the end of global recruitment.
  China Cohort: The China FAS included all randomized participants in the China cohort and were used for all China only efficacy analyses.
Time Frame: as for outcome 6
Population: Participants included in PD-L1-negative NSCLC and FAS analysis sets are reported in this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy | China: Durvalumab + Tremelimumab | China: SoC Chemotherapy
Number analyzed (Participants) | 410 | 413 | 78 | 82
months
  PD-L1-negative NSCLC analysis set: number analyzed (Participants) | 91 | 104 | 26 | 29
  PD-L1-negative NSCLC analysis set | 9.1 [6.9 to 12.8] | 12.4 [8.8 to 14.9] | 13.8 [10.1 to 27.4] | 10.3 [6.5 to 14.1]
  FAS | 9.4 [8.2 to 10.9] | 10.4 [9.1 to 11.5] | 15.5 [12.5 to 24.5] | 12.9 [9.2 to 15.4]
Statistical Analysis 1: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; PD-L1-negative analysis set: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab to be associated with a longer time to second progression than SoC; Test type: Superiority; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.748 to 1.388] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 2: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; PD-L1-negative analysis set: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab to be associated with a longer time to second progression than SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.360 to 1.219] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Global: Durvalumab + Tremelimumab vs Global: SoC Chemotherapy; FAS: Global: Durvalumab + Tremelimumab Vs Global: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab to be associated with a longer time to second progression than SoC; Test type: Superiority; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.845 to 1.147] — The HR and CI were calculated using a stratified Cox proportional hazards model, adjusting for PD-L1 status (>= 25% Vs < 25%), smoking status (never smoker Vs ever smoker) and histology (squamous Vs non-squamous), with ties handled by Efron approach
Statistical Analysis 4: Comparison: China: Durvalumab + Tremelimumab vs China: SoC Chemotherapy; FAS: China: Durvalumab + Tremelimumab Vs China: SoC Chemotherapy A HR <1 favors Durvalumab + Tremelimumab to be associated with a longer time to second progression than SoC; Test type: Other — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.492 to 1.030] — [estimate comment as in outcome 2, analysis 1]

15. Secondary Outcome: OS at Months 12, 18 and 24; Global Cohort: bTMB ≥20 Mut/Mb, bTMB ≥16 Mut/Mb, and bTMB ≥12 Mut/Mb Analysis Sets
Description: The OS was defined as the time from the date of randomization until death due to any cause (ie, date of death or censoring - date of randomization + 1).
  bTMB ≥20 mut/Mb, bTMB ≥16 mut/Mb and bTMB ≥12 mut/Mb analysis sets included the subset of participants in FAS whose bTMB status was ≥20 mut/Mb, ≥16 mut/Mb and ≥12 mut/Mb, respectively at baseline as defined by the GuardantOMNI CDx assay.
Time Frame: Months 12, 18 and 24
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy
Number analyzed (Participants) | 143 | 138
percentage of participants
  Month 12: bTMB ≥20 mut/Mb analysis set: number analyzed (Participants) | 69 | 60
  Month 12: bTMB ≥20 mut/Mb analysis set | 49.3 [37.1 to 60.4] | 40.8 [28.3 to 52.9]
  Month 12: bTMB ≥16 mut/Mb analysis set: number analyzed (Participants) | 93 | 89
  Month 12: bTMB ≥16 mut/Mb analysis set | 50.5 [40.0 to 60.2] | 48.9 [38.2 to 58.8]
  Month 12: bTMB ≥12 mut/Mb analysis set | 46.9 [38.5 to 54.8] | 44.6 [36.1 to 52.7]
  Month 18: bTMB ≥20 mut/Mb analysis set: number analyzed (Participants) | 69 | 60
  Month 18: bTMB ≥20 mut/Mb analysis set | 36.2 [25.1 to 47.4] | 20.4 [11.3 to 31.4]
  Month 18: bTMB ≥16 mut/Mb analysis set: number analyzed (Participants) | 93 | 89
  Month 18: bTMB ≥16 mut/Mb analysis set | 35.5 [25.9 to 45.1] | 28.5 [19.5 to 38.1]
  Month 18: bTMB ≥12 mut/Mb analysis set | 29.4 [22.1 to 36.9] | 27.8 [20.6 to 35.4]
  Month 24: bTMB ≥20 mut/Mb analysis set: number analyzed (Participants) | 69 | 60
  Month 24: bTMB ≥20 mut/Mb analysis set | 26.1 [16.4 to 36.8] | 13.6 [6.4 to 23.6]
  Month 24: bTMB ≥16 mut/Mb analysis set: number analyzed (Participants) | 93 | 89
  Month 24: bTMB ≥16 mut/Mb analysis set | 24.0 [15.8 to 33.2] | 18.2 [11.0 to 26.9]
  Month 24: bTMB ≥12 mut/Mb analysis set | 21.3 [15.0 to 28.4] | 19.0 [12.9 to 26.0]

16. Secondary Outcome: OS at Months 12, 18 and 24; Global and China Cohorts: PD-L1-Negative NSCLC and FAS Analysis Sets
Description: The OS was defined as the time from the date of randomization until death due to any cause (ie, date of death or censoring - date of randomization + 1).
  PD-L1-negative analysis set included the subset of participants in FAS whose PD-L1 status was PD-L1-negative at baseline as defined by the Ventana SP263 PD-L1 Assay (ie, <1% PD-L1-membrane expression in tumoral tissue).
  Global Cohort: The FAS included all randomized participants prior to the end of global recruitment.
  China Cohort: The China FAS included all randomized participants in the China cohort and were used for all China only efficacy analyses.
Time Frame: Months 12, 18 and 24
Population: Participants included in PD-L1-negative NSCLC and FAS analysis sets are reported in this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy | China: Durvalumab + Tremelimumab | China: SoC Chemotherapy
Number analyzed (Participants) | 410 | 413 | 78 | 82
percentage of participants
  Month 12: PD-L1-negative NSCLC analysis set: number analyzed (Participants) | 91 | 104 | 26 | 29
  Month 12: PD-L1-negative NSCLC analysis set | 47.8 [37.2 to 57.6] | 52.8 [42.6 to 61.9] | 68.0 [46.1 to 82.5] | 46.4 [27.6 to 63.3]
  Month 12: FAS | 47.7 [42.8 to 52.5] | 50.0 [45.0 to 54.8] | 72.8 [61.3 to 81.3] | 53.1 [41.7 to 63.2]
  Month 18: PD-L1-negative NSCLC analysis set: number analyzed (Participants) | 91 | 104 | 26 | 29
  Month 18: PD-L1-negative NSCLC analysis set | 34.1 [24.5 to 43.9] | 34.5 [25.4 to 43.8] | 44.0 [24.5 to 61.9] | 39.3 [21.7 to 56.5]
  Month 18: FAS | 34.8 [30.2 to 39.5] | 34.6 [30.0 to 39.3] | 54.6 [42.8 to 64.9] | 41.8 [31.0 to 52.3]
  Month 24: PD-L1-negative NSCLC analysis set: number analyzed (Participants) | 91 | 104 | 26 | 29
  Month 24: PD-L1-negative NSCLC analysis set | 22.1 [14.0 to 31.3] | 22.3 [14.7 to 30.9] | 36.0 [18.2 to 54.2] | 17.9 [6.5 to 33.7]
  Month 24: FAS | 25.7 [21.6 to 30.1] | 23.4 [19.4 to 27.7] | 44.2 [32.9 to 54.8] | 30.4 [20.7 to 40.6]

17. Secondary Outcome: Serum Concentrations of Durvalumab
Description: Blood samples were collected to determine the serum concentration of durvalumab.
Time Frame: Pre-dose and within 1 hour after end of infusion at Week 0 and 12; pre-dose on Week 24 and at follow-up Month 3
Population: Global Cohort: The FAS included all randomized participants prior to the end of global recruitment. Any participants recruited in China, after global recruitment had ended, were not included in the FAS.
  China Cohort: The China FAS included all randomized participants in the China cohort and were used for all China only efficacy analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | Global: Durvalumab + Tremelimumab | China: Durvalumab + Tremelimumab
Number analyzed (Participants) | 410 | 78
microgram per milliliter (µg/mL)
  Week 0: Pre-infusion: number analyzed (Participants) | 401 | 77
  Week 0: Pre-infusion | NA (NA) — NA = Below LLOQ. The LLOQ = 0.05 µg/mL. | NA (NA) — NA = Below lower limit of quantification (LLOQ). The LLOQ = 0.05 µg/mL.
  Week 0: End of infusion: number analyzed (Participants) | 399 | 76
  Week 0: End of infusion | 418.6 (74.8) | 392.7 (48.9)
  Week 12: Pre-infusion: number analyzed (Participants) | 239 | 52
  Week 12: Pre-infusion | 77.5 (138.1) | 72.4 (55.0)
  Week 12: End of infusion: number analyzed (Participants) | 236 | 52
  Week 12: End of infusion | 434.3 (105.6) | 448.9 (40.0)
  Week 24: Pre-infusion: number analyzed (Participants) | 129 | 35
  Week 24: Pre-infusion | 108.8 (95.7) | 85.6 (93.9)
  Follow-up Month 3: number analyzed (Participants) | 48 | 8
  Follow-up Month 3 | 8.8 (253.9) | 5.4 (351.7)

18. Secondary Outcome: Serum Concentrations of Tremelimumab
Description: Blood samples were collected to determine the serum concentration of tremelimumab.
Time Frame: Pre-dose and within 1 hour after end of infusion at Week 0 and 12, and at follow-up Month 3
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Global: Durvalumab + Tremelimumab | China: Durvalumab + Tremelimumab
Number analyzed (Participants) | 410 | 78
µg/mL
  Week 0: Pre-infusion: number analyzed (Participants) | 402 | 77
  Week 0: Pre-infusion | NA (NA) — NA = Below LLOQ. The LLOQ = 0.05 µg/mL. | NA (NA) — NA = Below LLOQ. The LLOQ = 0.05 µg/mL.
  Week 0: End of infusion: number analyzed (Participants) | 398 | 76
  Week 0: End of infusion | 20.3 (38.7) | 18.4 (43.3)
  Week 12: Pre-infusion: number analyzed (Participants) | 241 | 52
  Week 12: Pre-infusion | 3.4 (99.6) | 3.3 (64.6)
  Week 12: End of infusion: number analyzed (Participants) | 236 | 52
  Week 12: End of infusion | 20.8 (67.4) | 23.2 (43.4)
  Follow-up Month 3: number analyzed (Participants) | 46 | 11
  Follow-up Month 3 | NA (NA) — NA = Below LLOQ. The LLOQ = 0.05 µg/mL. | NA (NA) — NA = Below LLOQ. The LLOQ = 0.05 µg/mL.

19. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Response to Durvalumab
Description: Blood samples were measured for the presence of ADAs and ADA-neutralizing antibodies (nAb) for durvalumab using validated assays. ADA prevalence is defined as the percentage of participants with positive ADA result at any time, baseline or post-baseline. Treatment-emergent ADA is defined as the sum of treatment-induced ADA and treatment-boosted ADA. ADA incidence is the percentage of participants who were treatment-emergent ADA-positive. Treatment-boosted ADA is defined as baseline positive ADA titer that was boosted to >=4 fold during the study period. Persistently positive is defined as having at least 2 post baseline ADA positive measurements with at least 16 weeks (112 days) between the first and last positive measurements, or an ADA positive result at the last available assessment. Transiently positive is defined as having at least 1 post baseline ADA positive measurement and not fulfilling the conditions for persistently positive.
Time Frame: At Weeks 0, 12, and 24; 3 and 6 months after last dose of study treatment.
Population: Global Cohort: The FAS included all randomized participants prior to the end of global recruitment. Any participants recruited in China, after global recruitment had ended, were not included in the FAS.
  China Cohort: The China FAS included all randomized participants in the China cohort and were used for all China only efficacy analyses.
  The denominator for calculation of percentage for all categories is the number of ADA evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Global: Durvalumab + Tremelimumab | China: Durvalumab + Tremelimumab
Number analyzed (Participants) | 266 | 61
Participants
  ADA positive at any visit (ADA prevalence) | 26 | 1
  Treatment-emergent ADA positive (ADA incidence) | 12 | 1
  Treatment-boosted ADA | 0 | 0
  Treatment-induced ADA (positive post-baseline only) | 12 | 1
  ADA positive post-baseline and positive at baseline | 1 | 0
  Persistent positive | 11 | 1
  Transient positive | 2 | 0
  nAb positive at any visit | 3 | 0
  ADA positive at baseline and not detected post-baseline | 13 | 0

20. Secondary Outcome: Number of Participants With ADA Response to Tremelimumab
Description: Blood samples were measured for the presence of ADAs and ADA-nAb for tremelimumab using validated assays. ADA prevalence is defined as the percentage of participants with positive ADA result at any time, baseline or post-baseline. Treatment-emergent ADA is defined as the sum of treatment-induced ADA and treatment-boosted ADA. ADA incidence is the percentage of participants who were treatment-emergent ADA-positive. Treatment-boosted ADA is defined as baseline positive ADA titer that was boosted to >=4 fold during the study period. Persistently positive is defined as having at least 2 post baseline ADA positive measurements with at least 16 weeks (112 days) between the first and last positive measurements, or an ADA positive result at the last available assessment. Transiently positive is defined as having at least 1 post baseline ADA positive measurement and not fulfilling the conditions for persistently positive.
Time Frame: At Weeks 0 and 12; 3 and 6 months after last dose of study treatment.
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Global: Durvalumab + Tremelimumab | China: Durvalumab + Tremelimumab
Number analyzed (Participants) | 265 | 61
Participants
  ADA positive at any visit (ADA prevalence) | 49 | 2
  Treatment-emergent ADA positive (ADA incidence) | 37 | 1
  Treatment-boosted ADA | 1 | 0
  Treatment-induced ADA (positive post-baseline only) | 36 | 1
  ADA positive post-baseline and positive at baseline | 4 | 1
  Persistent positive | 29 | 0
  Transient positive | 11 | 2
  nAb positive at any visit | 33 | 0
  ADA positive at baseline and not detected post-baseline | 9 | 0

ADVERSE EVENTS:
Time Frame: Assessed until final analysis DCO for each cohort (24 June 2019 for Global Cohort and 21 September 2020 for China Cohort); maximum timeframe of approximately 44 months for each cohort.
Description: Global Cohort: The safety analysis set included all participants recruited prior to end of the global recruitment who received at least 1 dose of study treatment.
  China Cohort: The China safety analysis set included all participants recruited in the China cohort who received at least 1 dose of study treatment.
  All-Cause Mortality: Data from participants included in Global and China FAS was summarized separately. 30 participants in China cohort were also included in Global cohort.
Arm/Group | Global: Durvalumab + Tremelimumab | Global: SoC Chemotherapy | China: Durvalumab + Tremelimumab | China: SoC Chemotherapy
All-Cause Mortality (participants affected / at risk) | 328/410 | 329/413 | 50/78 | 62/82
Serious Adverse Events (participants affected / at risk) | 193/410 | 112/399 | 32/77 | 22/78
Other Adverse Events (participants affected / at risk) | 310/410 | 349/399 | 73/77 | 77/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global: Durvalumab + Tremelimumab (N=410) | Global: SoC Chemotherapy (N=399) | China: Durvalumab + Tremelimumab (N=77) | China: SoC Chemotherapy (N=78)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 11 (12) | 0 (0) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Haematotoxicity (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (6) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Optic neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 3 (3) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 4 (4) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 12 (12) | 1 (1) | 3 (3) | 0 (0)
Sudden death (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 27 (33) | 13 (15) | 3 (3) | 5 (6)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood calcium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood corticotrophin decreased (Investigations) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (8)
Platelet count decreased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraneoplastic arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Lateral medullary syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (3) | 3 (3) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (2) | 4 (4) | 2 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 1 (2) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 0 (0) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global: Durvalumab + Tremelimumab (N=410) | Global: SoC Chemotherapy (N=399) | China: Durvalumab + Tremelimumab (N=77) | China: SoC Chemotherapy (N=78)
Anaemia (Blood and lymphatic system disorders) | 59 (66) | 146 (201) | 25 (35) | 53 (74)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 38 (55) | 1 (1) | 13 (21)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 71 (113) | 2 (3) | 10 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (6) | 50 (73) | 0 (0) | 8 (11)
Hyperthyroidism (Endocrine disorders) | 34 (35) | 0 (0) | 9 (10) | 0 (0)
Hypothyroidism (Endocrine disorders) | 51 (58) | 2 (2) | 5 (12) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (7) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
Constipation (Gastrointestinal disorders) | 59 (64) | 84 (90) | 10 (13) | 9 (12)
Diarrhoea (Gastrointestinal disorders) | 72 (96) | 40 (53) | 5 (7) | 6 (7)
Nausea (Gastrointestinal disorders) | 57 (74) | 128 (244) | 10 (13) | 33 (108)
Stomatitis (Gastrointestinal disorders) | 9 (10) | 27 (40) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 29 (41) | 57 (80) | 8 (10) | 19 (34)
Asthenia (General disorders) | 50 (72) | 52 (59) | 9 (9) | 12 (16)
Fatigue (General disorders) | 56 (76) | 73 (95) | 1 (1) | 6 (9)
Malaise (General disorders) | 0 (0) | 0 (0) | 4 (4) | 7 (13)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 8 (9) | 5 (5)
Oedema peripheral (General disorders) | 29 (30) | 16 (23) | 6 (7) | 3 (3)
Pyrexia (General disorders) | 40 (51) | 32 (35) | 12 (21) | 9 (10)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Pneumonia (Infections and infestations) | 14 (14) | 20 (22) | 8 (9) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 6 (7) | 2 (2)
Alanine aminotransferase increased (Investigations) | 33 (39) | 34 (48) | 22 (27) | 22 (49)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 21 (34) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 27 (35) | 28 (41) | 25 (39) | 20 (38)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 4 (10) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 8 (12) | 2 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 6 (9) | 4 (6)
Blood creatinine increased (Investigations) | 8 (18) | 28 (36) | 0 (0) | 9 (12)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 8 (12) | 5 (5)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 3 (8) | 7 (8)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 4 (8) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 19 (33) | 10 (15)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 6 (9)
Lipase increased (Investigations) | 21 (30) | 7 (8) | 15 (26) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (10) | 29 (68) | 4 (8) | 35 (94)
Platelet count decreased (Investigations) | 2 (2) | 30 (51) | 3 (6) | 15 (30)
Weight decreased (Investigations) | 45 (46) | 16 (16) | 16 (16) | 4 (4)
Weight increased (Investigations) | 0 (0) | 0 (0) | 8 (10) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (9) | 35 (126)
Decreased appetite (Metabolism and nutrition disorders) | 69 (79) | 72 (88) | 14 (14) | 22 (37)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 11 (16) | 7 (10)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5) | 4 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (8) | 4 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 23 (31) | 15 (17)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (7) | 3 (3)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (13) | 7 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 13 (19) | 8 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (6) | 20 (24) | 5 (10) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 19 (38) | 15 (20)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (14) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 16 (19) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 (32) | 27 (53) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 29 (29) | 15 (15) | 7 (7) | 7 (16)
Dizziness (Nervous system disorders) | 20 (21) | 21 (21) | 4 (4) | 5 (6)
Headache (Nervous system disorders) | 24 (30) | 24 (25) | 5 (8) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 23 (28) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 22 (23) | 17 (18) | 5 (7) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (57) | 19 (22) | 11 (12) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 (33) | 16 (17) | 3 (3) | 6 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 10 (19) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 50 (50) | 0 (0) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 51 (62) | 11 (25) | 5 (5) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 58 (78) | 22 (25) | 12 (16) | 5 (6)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 7 (10) | 2 (2)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 4 (5) | 5 (18)

LIMITATIONS AND CAVEATS:
Analysis of the China cohort was performed to evaluate the consistency of efficacy and safety in Chinese participants with the global cohort in order to meet China health regulatory requirements and was not powered for a formal assessment of statistical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT02542293/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT02542293/SAP_001.pdf